CLINICAL TRIAL: NCT03261895
Title: Effectiveness of a Nurse-led Integrative Health and Wellness (NIHaW) Programme on Behavioural, Psychosocial and Biomedical Outcomes Among Individuals With Newly Diagnosed Type 2 Diabetes: A Randomised Controlled Trial
Brief Title: Effectiveness of a Nurse-led Integrative Health and Wellness Programme Among Newly Diagnosed Type 2 Diabetes Patients
Acronym: NIHaW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, YU Xingfeng, Graduate Assistant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NIHaW
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Nurse-led Integrative health and wellness programme
  Interventions: Behavioral: Nurse-led Integrative health and wellness programme
- control group (No Intervention): usual diabetes care

INTERVENTIONS:
Behavioral: Nurse-led Integrative health and wellness programme — Participants in the intervention group will go through a eight-session structured education programme. The education programme was designed by incorporating the evidences of diabetes care from the western medicine and the philosophy of traditional Chinese medicine.
  Arms: Intervention group

SUMMARY:
This randomized controlled trial aims to investigate the effectiveness of an integrative medicine (traditional Chinese medicine and western medicine) based structured education programme for newly diagnosed type 2 diabetes patients. The theoretical frame of this study is based on the health belief model and self efficacy theory. The hypotheses of this study are: 1) Participants in the intervention group will have higher level of self-management behaviour after intervention compared to participants in the control group; 2) Participants in the intervention group will have better diabetes knowledge after intervention compared to participants in the control group; 3) Participants in the intervention group will have higher level of self-efficacy after intervention compared to participants in the control group; 4) Participants in the intervention group will be less depressed after intervention compared to participants in the control group; 5) Participants in the intervention group will have better QOL after intervention compared to participants in the control group; 6) Participants in the intervention group will gain greater reduction in HbA1c after intervention compared to participants in the control group; 7) Participants in the intervention group will gain greater reduction in fasting blood glucose after intervention compared to participants in the control group; 8) Participants in the intervention group will gain greater reduction in BP after intervention compared to participants in the control group; 9) Participants in the intervention group will gain greater reduction in BMI after intervention compared to participants in the control group.

ELIGIBILITY:
Inclusion criteria:

* individuals diagnosed with type 2 diabetes in the preceding six months
* individuals aged ≥ 18 years
* individuals who were permanent residents of Xi'an City, China
* individuals without mental disorders
* individuals who were voluntary to participate in the study

Exclusion criteria:

* individuals with a terminal illness
* individuals who were physically disabled
* individuals who were taking part in other studies
* individuals with aural or visual problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Self-management | Baseline (T0)
  self-management refers to the efforts patients actively take to appropriately manage their daily life in order to gain optimal disease control, health status, and quality of life. Self-management was measured using the Summary of Diabetes Self-Care Activities (SDSCA) in this study.
Self-management | Immediately post-intervention (T1)
  self-management refers to the efforts patients actively take to appropriately manage their daily life in order to gain optimal disease control, health status, and quality of life. Self-management was measured using the Summary of Diabetes Self-Care Activities (SDSCA) in this study.
Self-management | Three months post-intervention (T2)
  self-management refers to the efforts patients actively take to appropriately manage their daily life in order to gain optimal disease control, health status, and quality of life. Self-management was measured using the Summary of Diabetes Self-Care Activities (SDSCA) in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Xingfeng YU, Principal Investigator — Chinese University of Hong Kong
Locations (4):
- China (4):
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Shaanxi Provincial People's Hospital, Xi'an
  - Xi'an Central Hospital, Xi'an

REFERENCES:
- [Derived] Yu X, Chau JPC, Huo L, Li X, Wang D, Wu H, Zhang Y. The effects of a nurse-led integrative medicine-based structured education program on self-management behaviors among individuals with newly diagnosed type 2 diabetes: a randomized controlled trial. BMC Nurs. 2022 Aug 5;21(1):217. doi: 10.1186/s12912-022-00970-7. PMID 35932073